CLINICAL TRIAL: NCT05637047
Title: Ultrasound-guided Pulsed Radiofrequency Versus Dry Needling for Pain Management in Chronic Neck and Shoulder Myofascial Pain Patients at a Tertiary Hospital in China: A Randomized Controlled Trial
Brief Title: Pulsed Radiofrequency vs Dry Needling in Myofascial Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Jin Wang, Doctor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRFversusDN
Record Dates: First submitted 2022-11-27; First posted 2022-12-05 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Myofascial Pain
MeSH Terms: interventions — Pulsed Radiofrequency Treatment; Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pulsed radiofrequency (Experimental)
  Interventions: Procedure: pulsed radiofrequency
- Dry needling (Active Comparator)
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Procedure: pulsed radiofrequency — ultrasound-guided intramuscular and interfascial pulsed radiofrequency ablation
  Arms: pulsed radiofrequency
Procedure: Dry needling — ultrasound-guided intramuscular and interfascial dry needling
  Arms: Dry needling

SUMMARY:
Myofascial pain (MPS) is the leading cause of chronic and persistent regional pain, affecting as many as 85% of the general population. A variety of treatment methods for myofascial pain have been investigated, including injection of saline, local anesthetics and steroids, dry needle, mini-scalpel, rich platelet plasma and radiofrequency ablation. Ultrasound guided dry needle (DN) and pulsed radiofrequency ablation (PRF) of the trigger point have been considered as two effective and promising treatments for myofascial pain. As far as searched, we failed to identify any study comparing the effects of DN and PRF in myofascial pain patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 70 years old.
2. Chronic (>3 months) myofascial pain in the neck, shoulder, and upper back region.
3. Myofascial pain will be diagnosed based on Simons and Travell's criteria: taut band palpable, exquisite spot tenderness of a nodule in a taut band, patient's recognition of current pain complaint by pressure on the tender nodule, and painful limit to full stretch range of motion.
4. Have at least a pain VAS score of 40 mm; thus, a minimal clinically significant change is detectable.

Exclusion Criteria:

1. History of receiving DN or PRF treatment or currently undergoing other pain-related treatments (acupuncture, laser, infrared therapy, etc.).
2. Presence or history of trauma, surgery, or infection in the pain region.
3. Current or history of taking moderate to strong analgesics, such as tramadol and morphine.
4. Severe systemic disease (eg. severe hepatic or renal dysfunction), coagulopathy, or medications affecting the coagulation system.
5. Allergy to medications used.
6. Pregnancy, psychiatric disease, medical background, inability to cooperate, or refusal to participate.

Withdrawn Criteria:

1. Unwilling to continue participation or unable to follow the treatment plan.
2. Unable to obtain the primary outcome data due to any reason.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain VAS score | Postoperative six months
  Pain evaluated by a 100mm line, 0mm indicates no pain, 100mm indicates the worst pain imaginable.

SECONDARY OUTCOMES:
Pain VAS score | postoperaitve day 0 and postoperative 1 and 3 months
  Pain evaluated by a 100mm line, 0mm indicates no pain, 100mm indicates the worst pain imaginable.
NDI | postoperaitve day 0 and postoperative 1, 3 and 6 months
  Neck disability index
PHQ9 | postoperaitve day 0 and postoperative 1, 3 and 6 months
  patient health questionnaire
GAD7 | postoperaitve day 0 and postoperative 1, 3 and 6 months
  generalized anxiety disorder (GAD-7) scale
Sleep status | postoperaitve day 0 and postoperative 1, 3 and 6 months
  Likert scale 1 to 5, 1 indicates very bad, 5 indicates very good
SF36 | postoperaitve day 0 and postoperative 1, 3 and 6 months
  health related quality of life short form 36 scale
Mechanical pain threshold | postoperaitve day 0 and postoperative 1, 3 and 6 months
  Mechanical pain threshold will be tested by pressing the pain point with an ergometer for three times and calculated the mean value of the pressure.

REFERENCES:
- [Derived] Wang J, Zhang Y, Cui X, Shen L. Ultrasound-guided pulsed radiofrequency versus dry needling for pain management in chronic neck and shoulder myofascial pain syndrome patients at a tertiary hospital in China: a randomised controlled trial protocol. BMJ Open. 2023 May 24;13(5):e071422. doi: 10.1136/bmjopen-2022-071422. PMID 37225266